CLINICAL TRIAL: NCT03948542
Title: Fractures of the Humeral Shaft With Primary Radial Nerve Palsy: Do Injury Mechanism, Fracture Type, or Treatment Influence Nerve Recovery: A Retrospective Study
Brief Title: Fractures of the Humeral Shaft With Primary Radial Nerve Palsy
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thomas Tiefenboeck, M.D., MSc, Principal Investigator, Medical University of Vienna
Other Study IDs: F.o.t.H. Version 1.0
Record Dates: First submitted 2019-03-19; First posted 2019-05-14 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Radial Nerve Palsy; Functional Outcome
Keywords: Intramedullary nailing; ORIF; Humeral shaft fracture
MeSH Terms: conditions — Radial Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Outcome: Nerve conduction studies (NCV) Functional assessment according to Daniels and Worthingham
  Interventions: Other: Outcome

INTERVENTIONS:
Other: Outcome — Nerve Recovery
  * NCV
  * Funcional assessment

SUMMARY:
This study addresses the question if patients with fractures of the humeral shaft and primary radial nerve palsy gain nerve recovery.

Additionally the influence of injury mechanism, fracture type, and treatment modality on nerve recovery should be evaluated.

DETAILED DESCRIPTION:
Adult fractures of the humeral shaft account for approximately 3% of all fractures; most can be treated nonoperatively. Due to the anatomy of the radial nerve and the entrapment between fragments in spiral fractures of the humerus, these injuries are associated with primary radial nerve palsy in up to 18%.

Therefore, the purpose of this study was to assess the influence of injury mechanism, fracture type, and type of surgical treatment on time to onset of nerve recovery and time to full nerve recovery in patients with humeral shaft fractures and concomitant primary radial nerve palsy.

A retrospective analysis of prospectively collected data for all patients treated with humeral shaft fracture and primary radial nerve palsy at an academic Level-I trauma center was performed. Between 1994 and 2013 a total of 615 patients with traumatic humeral shaft fractures were treated at the department. The dataset was examined for completeness and accuracy. Patients with an incomplete dataset, those with a pathologic or periprosthetic fracture, patients with non-surgical treatment, or who were younger than 18 years of age were excluded from this series. According to these criteria, a total of 50 patients with a humeral shaft fracture and primary radial nerve underwent surgical treatment

ELIGIBILITY:
Inclusion Criteria:

* patients treated with humeral shaft fracture and primary radial nerve palsy between 1994 and 2013 at the Department of Trauma Surgery, Medical University of Vienna
* surgical treatment
* complete data sets
* minimum 18 years of age

Exclusion Criteria:

* Patients with an incomplete dataset
* those with a pathologic or periprosthetic fracture
* patients with non-surgical treatment
* or who were younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include patients treated with humeral shaft fracture and primary radial nerve palsy between 1994 and 2013 at the Department of Trauma Surgery, Medical University of Vienna
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in nerve recovery; Nerve recovery after humeral shaft fracture and surgical treatment, Functional assessment | through study completion, from date of inclusion till first documented changes in nerve recovery, from date of admission assessed up to 36 months
  Functional assessment was routinely performed at all follow up visits including a clinical evaluation and muscle strength (M0-M5) with a manual muscle test that was graded according to Daniels and Worthingham.

SECONDARY OUTCOMES:
Nerve conduction studies (NCV) were performed routinely at two weeks following onset of radial nerve palsy and after 4 months in case of delayed recovery. | 2 weeks, 4 months
  Nerve conduction studies
Radiographic examination via X-ray in two planes | 3, 6 and 12 months after trauma
  X-ray in two planes

IPD SHARING:
Plan to Share IPD: No
Data will be available on request from the corresponding author in a blinded version